# TOPICAL USE OF VANCOMYCIN IN REDUCING STERNAL WOUND INFECTION IN CARDIAC SURGERY

## **Protocol**

Principal Investigator: Dr. John C. Mullen

Sponsored By University of Alberta

Protocol #: SWI-01-14

#### **GENERAL INFORMATION**

#### **PRINCIPAL INVESTIGATOR:**

Dr. John C. Mullen C/O Kayla-Marie Smith 2D2.18 WMC, 8440 112 Street Edmonton, AB, Canada T6G 2B7

Tel: (780) 966-8787

Email: akhani@ualberta.ca

#### **SPONSOR:**

The Governors of the University of Alberta 2-51 South Academic Building (SAB), University of Alberta Edmonton, AB, Canada T6G 2G7

Dr. Lorne Babiuk Vice President (Research)

Tel: 780-492-5353 / Fax: 780-492-3189

Email: lorne.babiuk@ualberta.ca

#### **CLINICAL CENTRE:**

University of Alberta Hospital / Mazankowski Alberta Heart Institute

#### **PROTOCOL DEVELOPMENT COMMITTEE:**

Abbas Khani-Hanjani, MD; Emily J Kuurstra, BSc

## **TABLE OF CONTENTS**

| TABLE OF CONTENTS | 3 |
|--------------------------------------------------|----|
| STUDY SUMMARY | 4 |
| DATA COLLECTION SUMMARY | 5 |
| ABREVIATIONS & ACRONYMS | 6 |
| BACKGROUND | 7 |
| OBJECTIVES | 7 |
| TRIAL DESIGN | 7 |
| TREATMENT ASSIGNMENT | 7 |
| RANDOMIZATION | 8 |
| MASKING | 8 |
| INVERVENTIONAL AGENT | 8 |
| ELIGIBILITY CRITERIA | 9 |
| DATA COLLECTION | 9 |
| ENDPOINTS | 10 |
| ADVERSE EVENTS | 11 |
| DATA MANAGEMENT | 11 |
| STATISTICAL ANALYSIS | 11 |
| PLANTRIAL CONDUCT | 12 |
| REFERENCES | 13 |
| APPENDIX I: CARDIAC SURGERY DATA COLLECTION FORM | 14 |

| APPENDIX II: SURGICAL SITE INFECTION SURVEILLANCE FORM | 19 |
|--------------------------------------------------------|----|
| APPENDIX III: CASE REPORT FORMS | 22 |

## **STUDY SUMMARY**

| Title | Topical Use of vancomycin in Reducing Sternal Wound Infection in Cardiac Surgery |
|---|---|
| Objective | To determine if using topical vancomycin as a prophylactic treatment during open heart surgery will reduce the incidence of sternal wound infection (SWI). |
| Methodology | Prospective, double-blind, randomized (1:1) controlled trial. |
| Rx Arms | During open heart surgery, patients will have a 4x8 inch piece of sterile gauze covering each side of the divided sternum. The gauze will be soaked in the following solutions: Group 1: 5 g vancomycin dissolved in 50 mL sterile water for injection Group 2: 50 mL sterile water for injection |
| Number of Subjects | A total of 1,552 patients will be randomized to either vancomycin or no vancomycin. This will provide an 80% power to detect a 50% reduction in infection rates (7% versus 3.5%). |
| 1° Endpoints | The incidence of SWI (including superficial incisional, deep incisional, and organ/space surgical site infections) at 3 months postoperative. |
| 2° Endpoints | <ul> <li>Incidence of SWI at 1 year postoperative</li> <li>Duration of index hospitalization and subsequent readmissions due to SWI</li> <li>Use of prophylactic antibiotics</li> <li>Cost analysis</li> <li>Adverse events</li> </ul> |
| Duration | Accrual is expected to take 3 years. All patients will be followed for one year postoperatively. |
| Inclusion Criteria | <ul> <li>Able to sign Informed Consent and Release of Medical Information Form</li> <li>Age ≥ 18 years</li> <li>Undergoing cardiac surgery with complete sternotomy (including reoperations)</li> </ul> |
| Exclusion Criteria | <ul> <li>Evidence of active infection (any culture positive or blood positive infection)</li> <li>Undergoing organ transplantation</li> <li>Patients with known hypersensitivity to vancomycin</li> <li>Pregnant or nursing women</li> <li>Mental impairment or other conditions that may not allow participant to understand the nature, significance, and scope of study</li> </ul> |

## **DATA COLLECTION SUMMARY**

| ASSESSMENT | BASELINE | PROCEDURE | PRE-DISCHARGE | EVENT DRIVEN |
|---|---|---|---|---|
| Informed Consent | X | | | |
| Eligibility and Enrollment | Χ | | | |
| Baseline Characteristics | X | | | |
| Index Surgery | | X | | |
| Index Hospital Discharge | | | X | |
| Postoperative Laboratory Results | | | X | Х |
| APPROACH Data | X | X | X | X |
| ProvServ Data | | | X | X |

## **ABBREVIATIONS & ACRONYMS**

| SWI | Sternal wound infection |
|---|---|
| DM | Diabetes mellitus |
| OR | Operating room |
| EPICORE | Epidemiology Coordinating and Research |
| DIN | Drug Identification Number |
| APPROACH | Alberta provincial project for outcome assessment in coronary heart disease |
| RedCap | Research electronic data capture |
| CR | Creatinine |
| GFR | Glomerular filtration rate |
| QMCR | Quality management in clinical research |
| HREB | Health research ethics board |
| HGB | Hemoglobin |
| HCT | Hematocrit |
| PLT | Platelet count |
| WBC | White blood cell count |
| NEUT | Neutrophil count |
| LYMPH | Lymphocyte count |
| MONO | Monocyte count |
| EOS | Eosinophil count |
| BASO | Basophil count |
| Na | Sodium |
| K | Potassium |

#### **BACKGROUND**

Sternal wound infection (SWI) is an uncommon yet serious risk associated with open heart surgery. Both superficial and deep SWI are associated with significant comorbidities, longer hospital stay and costs. Deep SWI affects 1-3% of patients postoperatively with a mortality rate of 20-30% for patients who develop mediastinitis [1-3]. A number of risk factors – such as diabetes (DM), obesity, and complex cardiovascular operations requiring longer surgical time – have been associated with the development of SWI [1]. Given that these risk factors are on the rise in today's cardiovascular surgical practices, alternative strategies should be considered to reduce and/or avoid the complication of SWI. Topical use of antibiotics has been shown to be effective in reducing at least Deep SWI both in small randomized studies and Meta analyses [3-4]. The most common bacterial culprits in SWI are staphylococcus species that are mostly sensitive to Vancomycin. However, systemic use of these antibiotics is associated with drug side effects such as nephrotoxicity and therefore their use is limited in patients with renal failure or insufficiency, which make up a significant number of patients undergoing open heart surgery. Studies have shown that the use of topical Vancomycin could be both safe and effective in reducing deep SWI even in patients with renal failure and insufficiency [5, 6]. Vancomycin is currently being used topically in a number of American centres (such as Cleveland Clinic and Boston Medical Center [5]). However, the topical use of vancomycin is considered off-label use of this drug in Canada and is not generally being used. The current overall rate of superficial and deep SWI in our institute is around 7%, the proposed study will attempt to assess and reduce the rate of SWI in patient undergoing open heart surgery.

#### **OBJECTIVES**

The primary objective of this clinical trial is to determine if using topical vancomycin as a prophylactic treatment during open heart surgery will reduce the incidence of SWI.

#### **TRIAL DESIGN**

This is a double-blind, randomized clinical trial. The study will be conducted at the University of Alberta Hospital and 1,552 patients will be randomized. All patients will be followed for one year postoperatively.

#### TREATMENT ASSIGNMENT

During open heart surgery, patients will have one piece of sterile gauze covering each side of the divided sternum. The investigators intend to use Derma Sciences Inc. Dupaque X-Ray Detectable 4 x 8 inch sponges for the purpose of this study. The gauze will be soaked in one of the following solutions (depending on the randomized treatment assignment) until the solution is absorbed (approximately 1-2 minutes):

Group 1: 5 g vancomycin dissolved in 50 mL sterile water for injection

Group 2: 50 mL sterile water for injection

The soaked gauzes will be applied and remain on the divided sternum once hemostasis has been achieved. The gauzes will be removed in the operating room (OR) at the end of the surgical procedure(s), just prior to chest closure.

#### **RANDOMIZATION**

Patients will be randomized in a 1:1 fashion. By this arrangement, 50% of the patients will receive topical vancomycin (Group 1) and 50% will not receive topical vancomycin (Group 2) during open heart surgery.

#### **MASKING**

This is a double-blind, sham procedure controlled trial. In order to maintain blinding of the investigators, the study coordinators, and the patients, Epidemiology Coordinating and Research (EPICORE) Centre will create a confidential randomization key. This key will be provided to the site's Research Pharmacy Office in order to guide the preparation of masked syringes containing either 5 g vancomycin dissolved in 50 mL sterile water (Group 1) or 50 mL sterile water (Group 2). The syringes will be prepared in small batches and labeled with expiration dates based on the chemical stability (96 hours) of vancomycin in sterile water for injection at a concentration of 100 mg/mL [7]. The study syringes will be stored in a refrigerator in the OR and therefore readily available for use.

#### INTERVENTIONAL AGENT

The interventional agent to be used in this clinical trial is <sup>Pr</sup>vancomycin hydrochloride for injection, USP (Pharmaceutical Partners of Canada Inc, Richmond Hill, ON). The product's Drug Identification Number (DIN) is 02139383.

#### **ADVERSE REACTIONS**

There have been rare reports of renal failure in patients treated intravenously with vancomycin, particularly when given large doses [7]. Most of these cases involved patients who had pre-existing kidney dysfunction or patients who received concomitant aminoglycosides.

The development of reversible neutropenia has been reported; usually beginning at least a week after the onset of treatment with vancomycin or after a total dose of more than 25 g has been administered [7].

Approximately two dozen patients have reported hearing loss associated with the use of vancomycin [7]. In most of these cases, patients also had kidney dysfunction, pre-existing hearing loss, or concomitant treatment with an ototoxic drug.

#### **DOSE RATIONALE**

Topical use of 5 g of vancomycin, in paste form, has been shown to reduce the rate of deep SWI without any significant adverse effect on the patient undergoing open heart surgery [5]. However there is no double blinded randomized controlled study to confirm the effectiveness of topical vancomycin in reducing SWI. The current randomized controlled trial will use 5 g of solubilized vancomycin, in 50 mL of sterile water for injection, for a topical application on sternal wound to evaluate the rate of total sternal wound (superficial and deep) infection.

07-May-2019

Note: The investigators intend to use Sterile Water for Injection USP (Baxter Corporation, Mississauga, ON) based on availability (DIN: 02014882).

#### **ELIGIBILITY CRITERIA**

#### **INCLUSION CRITERIA**

- Able to sign Informed Consent and Release of Medical Information Form
- Age ≥ 18 years
- Undergoing cardiac surgery with complete sternotomy (including re-operations)

#### **EXCLUSION CRITERIA**

- Evidence of active infection (any culture positive or blood positive infection)
- Undergoing organ transplantation
- Patients with known hypersensitivity to vancomycin
- Pregnant or nursing women
- Mental impairment or other conditions that may not allow participant to understand the nature, significance, and scope of study

#### **DATA COLLECTION**

The majority of data collected in this trial will be obtained from pre-existing hospital databases. The Alberta Provincial Project for Outcome Assessment in Coronary Heart Disease (APPROACH) database will be the source of information such as the patients' medical history, index procedure, and in-hospital postoperative complications. The Cardiac Surgery Data Collection Form (APPENDIX I) contains a complete list of data elements that will be obtained from the APPROACH database.

Alberta Health Services' ProvServ database maintains record of all patients who are treated at the clinical site for SWI, within one year of surgery. This database will provide follow-up information regarding the incidence of SWI in both study groups. A complete list of data elements that will be obtained from the ProvServ database can be found on the Surgical Site Infection Surveillance Form (APPENDIX II).

All data collected using the Case Report Forms (APPENDIX III) will be entered into the Research Electronic Data Capture (REDCap) system created by EPICORE Centre.

#### **CONSENT**

Prior to protocol-defined data collection, the study personnel will meet with the potential study participant to thoroughly discuss the nature of the clinical trial. All risks and benefits of the study will be explained; and all questions will be answered to the satisfaction of the participant prior to signing the informed consent form.

#### **ELIGIBILITY AND ENROLLMENT**

The inclusion and exclusion criteria will be document by the study personnel prior to randomization. All consented patients will be given a unique 5-digit identification code which will be used throughout the course of the study.

#### **BASELINE CHARACTERISTICS FORM**

This form captures the necessary patient identifiers that will be used to match and pull data from the hospital's databases. Information pertaining to the patient's baseline functionality, immune system functionality, and laboratory results will also be collected. The study personnel will obtain laboratory results from routine preoperative blood work, specifically selecting the assessment that was performed closed to the patient's index surgery.

#### **INDEX SURGERY FORM**

The identification number of the used masked syringes will be recorded, as well as any adverse reactions to the study product observed within 24 hours.

#### **INDEX HOSPITAL DISCHARGE FORM**

This form captures whether the patient is discharged on antibiotic medications.

#### **POSTOP LABORATORY RESULTS FORM**

The study personnel will review the standard of care postoperative laboratory results listed on this form and record the last value obtained for each parameter, prior to index hospital discharge. If the creatinine (CR), or Glomerular filtration rate (GFR) is abnormal at this time, the patient's laboratory results will be monitored post-hospital discharge. The study personnel will record all protocol-defined laboratory results until the patient has reached their baseline value (± 10%) or normal range; or until they have reached one year postoperative (whichever comes first).

#### **ENDPOINTS**

#### **PRIMARY ENDPOINTS**

#### Incidence of SWI

The primary endpoint of this trial is the incidence of SWI at 3 months postoperative. This includes superficial incisional, deep incisional, and organ/space surgical site infections as defined in Appendix II. The data will be obtained from the ProvServ database.

#### **SECONDARY ENDPOINTS**

#### Incidence of SWI

The incidence of SWI at 1 year postoperative will also be determined.

#### <u>Duration of index hospitalization and subsequent re-admissions due to SWI</u>

The length of hospital stay from index surgery to hospital discharge will be recorded for all patients. The duration of subsequent re-admissions due to SWI will also be documented.

#### Use of prophylactic antibiotics

The use of prophylactic antibiotics at index hospital discharge will be recorded for all patients. The ProvServ database will also provide information regarding the use of prophylactic antibiotics for those patients returning to hospital with signs of infection.

#### Cost analysis for SWI treatment

The study personnel will obtain hospital costing data for the various assessments and procedures involved in the treatment of SWI. This will allow comparisons to be made regarding the cost effectiveness of using topical vancomycin as a prophylactic treatment.

#### Adverse events

The study personnel will document and compare the occurrence of adverse events in each treatment group (see the Adverse Events section for further details).

#### **ADVERSE EVENTS**

#### RENAL INSUFFICIENCY/FAILURE

Defined as significant increases in creatinine or decreases in glomerular filtration rate between baseline and pre-discharge laboratory results.

#### **N**EUTROPENIA

Abnormally low postoperative neutrophil count.

#### **HEARING LOSS**

New onset hearing loss or worsening of a pre-existing condition.

#### **ALLERGIC REACTIONS TO VANCOMYCIN**

Abnormal redness or sensitivity of skin at the site of vancomycin application. Hypotension following the administration of vancomycin.

#### **GENERAL**

Further postoperative complications/adverse events will be obtained from the APPROACH database. Please refer to APPENDIX I for a complete list.

#### **DATA MANAGEMENT**

All study data actively collected by the study personnel (APPENDIX III) will be entered in the secure web-based REDCap system. Study personnel requiring access will have their own login and password. Data obtained from the hospital databases (APPENDICES II-III) will be collected and stored according to the security measures currently implemented by the custodians of the databases.

On-site monitoring will be provided by the University of Alberta's Quality Management in Clinical Research (QMCR), as per established guidelines.

#### STATISTICAL ANALYSIS PLAN

The statistical plan and analysis for this study is being provided by EPICORE Centre.

#### **ANALYSIS OF PRIMARY END POINT:**

The primary analysis will compare the proportions of patients having sternal wound infection between the two treatment groups using chi-squared test. Analyses will be performed according to the intention-to-treat principle. Descriptive statistics including frequency distributions, percentages, means and standard deviations will be presented for the baseline variables. The median and the IQR (Inter Quartile Range) will be used to represent variables with skewed distributions. The baseline variables will be compared between the treatment groups using chi-squared test, t-test or Wilcoxon Mann-Whitney test, as appropriate. If necessary, a multi-variable analysis will be performed using logistic regression to control potential confounding effect in the analysis stage. All the statistical tests will be two-sided. A p-value of <0.05 will be considered statistically significant.

#### **ANALYSIS OF SECONDARY END POINTS:**

Secondary end points will be evaluated at the end of the study. Duration of index hospitalization between the treatment groups will be compared using survival analysis. The log rank test will be used. The total and the mean number of readmissions between the two groups will be compared by t-test or Wilcoxon Mann-Whitney test, as appropriate. A chi-squared test will be used to compare the use of prophylactic antibiotics. Cost analysis will be performed by comparing means or medians between the groups using t-test or Wilcoxon Mann-Whitney test, as appropriate. If necessary, multi-variable linear or logistic regression will be performed for the secondary end points, as appropriate. All the statistical tests will be two-sided. A p-value of <0.05 will be considered statistically significant.

#### **ANALYSIS OF ADVERSE EVENTS:**

Adverse events will be reported by frequency tables, percentages, means, standard deviations, medians or IQRs as appropriate at the interim and the final analysis. Proportions of adverse events between the groups will be compared by chi-squared test. Means or medians will be compared by t-test or Wilcoxon Mann-Whitney test, as appropriate. Count data will be compared by Poisson regression.

#### **INTERIM ANALYSIS:**

One interim analysis will be performed in a half way of the trial (after 776 patients will be followed). Interim analysis will be performed on the primary end point and the adverse events using a two-sided significance test with O'Brien-Fleming type spending function and a type I error rate of 5%.

#### TRIAL CONDUCT

This study will be conducted in compliance with the protocol approved by the University of Alberta Health Research Ethics Board (HREB), and according to Good Clinical Practice standards. No deviation from the protocol will be implemented without the prior review and approval of the HREB except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the HREB as soon as possible.

#### **REFERENCES**

- [1] Borger MA, Rao V, Weisel RD, et al. Deep sternal wound infection: risk factors and outcomes. Ann Thorac Surg 1998;65:1050-6.
- [2] Mauermann WJ, Sampathkurmar P, Thompson RL. Sternal wound infections. Best Pract Res Clin Anaesthesiol 2008;22:423-36.
- [3] Friberg O, Svedjeholm R, Söderquist B, Granfeldt H, Vikerfors T, Källman J. Local gentamicin reduces sternal wound infections after cardiac surgery: a randomized controlled trial. Ann Thorac Surg 2005;79:153-61.
- [4] Mavros MN, Mitsikostas PK, Alexiou VG, Peppas G, Falagas ME. Gentamicin collagen sponges for the prevention of sternal wound infection: A meta-analysis of randomized controlled trials. J Thorac Cardiovasc Surg 2012;144:1235-40.
- [5] Lazar HL, Barlam T, Cabral H. The effect of topical vancomycin applied to sternotomy incisions on postoperative serum vancomycin levels. J Card Surg 2011;26:461-5.
- [6] Vander Salm TJ, Okike ON, Pasque MK, Pezzella AT, Lew R, Traina V, Mathieu R. Reduction of Sternal Infection by Application of Topical Vancomycin. Thorac Cardiovasc Surg 1989;98:618-22.
- [7] Pharmaceutical Partners of Canada Inc., Product Monograph, PrVANCOMYCIN HYDROCHLORIDE FOR INJECTION, USP. Control # 144773, March 7, 2011.

## **APPENDIX I: CARDIAC SURGERY DATA COLLECTION FORM**





## Cardiac Surgery Data Collection Form

| Case Number 2014 | Patient Medical Reco | ord |
|---|---|---|
| Last Name: | First Name: | MI |
| Ht:kg OR S | Start date/time | End Time |
| Surgeon: Re | esident: | Anesthetist: |
| CCS: NYHA: Su<br>Diseased Vessels: Le | rgery Type:<br>ft Main: YesNo Most Re | sp Diagnosis |
| Operative Procedure: | | |
| ☐Aortic Dissection ☐Acute | ☐TMLR ☐DOR ☐ ☐Tumor ☐Transpla ☐Asc w/o root ☐Arch ☐Des ☐Abd-infra ☐AAA Endo ☐AAA ☐Chronic ☐Type A ☐Typ | e B |
| ☐ Other Non-Cardiac ☐ Carotid Endar☐ ☐ Fem-fem Bypt☐ ☐ Lung Transplant ☐ Type L R B | terectomy | horacic |
| Incidence: □1 <sup>st</sup> Op □Reop 1 <sup>st</sup> , If Reop is it Same Adm? Angina (72 Hr) Tracking Adm d/t | 2 <sup>nd</sup> , 3 <sup>rd</sup> , 4 <sup>th</sup> , Reason fo<br>Unique Record Yes/No Old R | or Reop:<br>ecord #<br>To Unit |
| □CABG □Valve Replace □A □M □T □P □Valve Repair □A □M □T □P □Aortic Aneurysm □Asc+Root □Abd-supra □Aortic Dissection □Acute □Other Non-Cardiac □Carotid Endal | Other LVA Septal M Cardiac Congenital ASD TMLR DOR Tumor Transplate Asc w/o root Arch Destended Abd-infra AAA Endo AAA Chronic Type A Type Type A Type Type A Asc Chronic Asc Chronic Asc Chronic As | □VSD □Maze □Atrial Ablation □Trauma □Bental □Aortic Repair ant □Other □ Sc □Thoracic A open □TAA □ De B □Thoracic □Other □ De |
| Indication/Cardiac Status (if ACS get Selection Factors LVEF% Calc / Est by LVEDPmm Angio | Outcome Determinants Hypertension Hyperlipidemia mmol/L CholTG | Prior Infarction D/T<br>Prior PCI<br>Prior CABG<br>Congestive Heart Failure |
| Mean PAP | HDLLDL Renal Failure | PAD / PVD Cerebrovascular Disease -Type Infective Endocard |

| ☐ Digitalls ☐ ☐ Coumadin ☐ ☐ Inotropes ☐ ☐ Steroids ☐ ☐ | Nitrates IV Diuretics Oral Hypoglycemic Anticoagulants – I Gly IIb IIIa Inhib – Lipid Lowering – s | ⊟A<br>: □III<br>Heparir<br>Abcixin | ı (Uı<br>nab | (As<br>in<br>nfra<br>(Re | piri<br>c/l\<br>oPi | n)<br>/)/ | [<br>He | □AD<br>□Am<br>parin | B Inhibitors<br>P Inhib – Clopidogi<br>ilodarone<br>(Low molec.) / Thr<br>itied (Integrilin) / Til | ombin inhibitors |
|---|---|---|---|---|---|---|---|---|---|---|
| Bypass Data: Endarterectomy Perform Arterioplasty: Yes/No # of Dist Anast with Very of Dist Anast with Arterioplasty in the Arteriop Graft Revision: Prior PCI Vessels: | nous:<br>terial: | | f IN | ΛA | Dis | stal | : | ifts:_<br>No | | st site: |
| Diseased Vessels: LN CXOM1 Vessels Grafted: LN CXOM1 | OM2OM3 | 11 | D2<br>D2 | RO | ĒΑ | 3_ | _^ | RI_<br>M_<br>RI_<br>M_ | PDACB_ | <del></del> |
| Valve Data: Dx St<br>Aortic<br>Mitral<br>Tricuspid<br>Pulmonary | enosis Insu | | Etiol | logy | у<br> | | | 100 | Gradient ( | Cath/Echommhgmmhgmmhgmmhg |
| Valve Surgery: Actic Procedure: No Replacement Repai/Reconstruction Root Reconstruction w/ Valve Cor Replacement + Actic Graft Conde Root Reconstruction av/ Valve W/ Replacement Actic Valve w/ Replacement Accending Act Replacement Accending Act Replacement Accending Act Replacement Accending Act Resection Sub-Actic Stancels | ring (if Replacement Mitral Repair Attr | (Annulop<br>(é Annulo<br>ni) | plasi | ty | | No<br>Ann<br>Rep<br>Rec | ulos<br>ince<br>onsi | ruction | | Pulmonic Procedure No Replacement Reconstruction |
| Aortic Annular Enlargement: Yes<br>↓ Key M = Mechanical B = B | ioprostresis H = Hom | | | = Au | - | | | | R = Ring/Annuloplasty | BA = Band/Annulophesty Size:(mm) |
| Aortic Prosthasis - | Implant Type: | None | | | | | | BA | Explant: | W. S. S. |
| | Explant Type: | None | 1.4 | | | A | (2020) | BA | | Size:(mm) |
| Mitral Prosthesis - | Implant Type: | None | | | | | | BA | | Size:(mm) |
| | Explant Type: | None | | | | | | BA | The second second | Size:(mm) |
| Tricuspid Prosthesis - | Implant Type: | None | | | 200 | | | BA | | Size:(mm) |
| | Explant Type: | None<br>None | | | | | | BA | * | - C 4.55 may |
| Pulmonic Prosthesis - | implant Type:<br>Explant Type: | None | | 250 | | | | | * G.F. 17 17 17 18 | Size:(mm) |

Mazankowski Alberta Heart Institute

08/20/13

2

| <b>CPB Data</b><br>OH# 14 <u>-</u> | _ Perfusionist: | X( | Clamp | min Pump | min |
|---|---|---|---|---|---|
| On Pump Case Ye | s/No | If No X | Clamp, give | reason | |
| Cardioplegia Yes/N | No Co | onversion from off pur | mp to on pum | p Yes/No | |
| Low Core Temp | Pre-o | p HgB | Pre-pump Ho | gB | |
| Ordered or | Given Prior to Surge | ery Yes/No<br>of incision Yes/No<br>ostop (post surgical er | (within 2 hrs<br>nd time) | if Vanco or Fluoroq<br>Yes/No | uinolone) |
| Intraop Medication | s | sylol 🔲 Tran | examic Acid | | |
| Cannulation Metho | d Arterial: ☐Femo<br>Venous: ☐Femo | oral ∐Arch ∐Aso<br>oral ∐Jugular ∏/ | c Aorta 🔲 Atrial (2 stage | OtherBio | caval |
| IABP Yes/No Tim<br>VAD Yes/No Tim | inging | _Reason<br>_Type | | | |
| Intraop TEE Yes/<br>Inotropes Leaving | | eturn to CPB Yes/No<br>ntiarrhythmics Leavin | o if Yes: On<br>ig OR Yes/N | ce More than One | ce |
| Blood Products (# | of units)<br>a-op | Post-op | | | |
| RBC | | | | | |
| Cryo<br>Platelets | | | | | |
| Postop Studies wi<br>ECHO Yes/No | thin 30 Days Y<br>Cath Yes/No | es/No<br>PCI Yes/No | Other | | |
| First Extubation D | | Time:<br>'es/No | | | |
| Reintubation Durin | 19 1 100 7 1 1 1 1 1 | | | | |
| | te: | _ Time: | | | |
| The state of the s | te: | _ Time: | | | |
| Reintubation Da | te: | Time: | | | |
| Extubation Da | te: | Time: | | | |
| | te: | Time:<br>Time: | | | |
| Extubation Da | te: | | | | |

| Postop Com | plications: Yes/No If Yes: <30 Days >30Days |
|---|---|
| Pulmonary: | Yes/No |
| | ☐ Prolonged Vent ☐ Pulm Embolism ☐ Pneumonia ☐ ARDS |
| | ☐ Chest Tube ☐ Pulm Edema ☐ Pleural Effusion ☐ Pneumothorax |
| Reoperation: | Yes/No |
| | ☐Bleeding ☐Graft Occlusion ☐Other Non-Cardiac ☐Valve Dysfunction |
| | Uther Cardiac Reop Date Type Surg |
| | Reop Date lype Surg |
| Neurologic: | Yes/No |
| | Postop Stroke for > 72 hrs |
| 1-51' | ☐Continuous Coma >=24 hrs ☐Paralysis ☐Other |
| Infection: | Yes/No |
| Panel. | ☐Sternum Super/Deep ☐Thoracotomy ☐Arm ☐Leg ☐Septicemia |
| Renai: | Yes/No Postop Creatinine Level (Peak) |
| Vascular: | If Yes is Dialysis Required? Type: Prisma or Hemo or Both |
| Cardiac: | ☐Illiac/Femoral Dissection ☐Acute Limb Ischemia Yes/No |
| Cardiac. | ☐Peri-op MI ☐Heart Block ☐Cardiac Arrest ☐Atrial Fib ☐VT/VFib |
| | □Low CO □Bradycardia □Tamponade □Anticoag Comp |
| | Other |
| Gastrointestina | al: Yes/No |
| | ☐ Ischemia ☐ Gl Surgery ☐ Other |
| CV ICU Readr | mission: Yes/No |
| | Imission Reason If "Other" |
| Discharge State | tus: Home Other Facility Extended/Transitional Care/Rehab |
| | Nursing Home Deceased To OR for Re-op Unknown |
| <b>.</b> | |
| Discharge Date | e/Time: |
| Potogral: | Cardina Bahahilitatian Van/No Antinanalatian Ott to Antinanalatian |
| Neienal. | Cardiac Rehabilitation: Yes/No Anticoagulation Clinic: Yes/No |
| Cause of Deat | h: Primary COD: |
| Cardia | |
| Vascula | |
| , door | ar Fairaiai Caici Circiowii |
| Readmission w | vithin 30 Days: Yes/No |
| Primary | Reason |
| Second | lary Reason |
| Procedi | ure Done |
| Discharge Med | ls: Transplant Meds Given: |
| | ☐ Solu-medrol |
| ☐ Beta Blockers ☐ Lipid Lowering - Statin / Non-Statin ☐ ATGAM / RATGAM | |
| ☐ ACE Inhibitors ☐ ASA (Aspirin) ☐ Zenapax / Daclizumab | |
| ADP Inhibitors Antiamhythmics - Amiodarone / Other Basiliximab | |
| □ARB | Inhibitors |
| | Cyclosporine |
| | ☐ MMF / CellCept |
| | ☐ Prednisone |

Mazankowski Alberta Heart Institute

01/14/14

4

## **APPENDIX II: SURGICAL SITE INFECTION SURVEILLANCE FORM**



| Name | _ |
|--------------|---|
| AB PHN/ULI | _ |
| Hospital ID# | _ |

## Surgical Site Infection Surveillance Form

| Revised: May 2014 for UAH & Stollery | |
|---|---|
| | DEMOGRAPHIC DATA |
| Name: | |
| Last name First Name | Middle Name |
| Date of Birth: | Gender: AB PHN/ULI: |
| (yyyy/mmm/dd)/ | ☐ M ☐ F ☐ Unk |
| Hospital ID # Unk | CHEC # (if applicable) |
| <u> </u> | , , , , |
| Procedure Type: | RGICAL INFORMATION Bilateral Procedure: |
| Provincial-Total Hip Replacement (TH) | Bilateral Procedure. Y N Dollor Site. |
| Provincial-Total Knee Replacement (TK) | Right |
| Other: (see reverse) | Left |
| Procedure Date: | Incision Start Time: |
| (yyyy/mmm/dd)/ | Incision Closure Time & Date: |
| Classification: Clean Clean-Contaminated | |
| ☐ Contaminated ☐ Dirty-Infected | <b>ASA Score</b> : □ 1 □ 2 □ 3 □ 4 □ 5 |
| Procedure Zone: | Procedure Facility: |
| Name of Surgeon: | |
| Antibiotic Prophylaxis Acceptable Unacceptable | Antibiotic Prophylaxis Re-dose Acceptable Unacceptable |
| ☐ Unable to collect | ☐ Unable to collect |
| ☐ None Given | ☐ None Given |
| ☐ Cefazolin (ancef) ☐ 1g ☐ 2g | ☐ Cefazolin (ancef) ☐ 1g ☐ 2g |
| ☐ Ciprofloxacin ☐ 400 mg | ☐ Ciprofloxacin ☐ 400 mg |
| ☐ Clindamycin ☐ 600mg ☐ 900mg | ☐ Clindamycin ☐ 600mg ☐ 900mg |
| ☐ Flagyl ☐ 500 mg | ☐ Flagyl ☐ 500 mg |
| ☐ Gentamicin ☐ 7 mg/kg | ☐ Gentamicin ☐ 7 mg/kg |
| │ | ☐ Vancomycin ☐ 1g ☐ 1.5g |
| Other (specify): | ☐ Other (specify): |
| Antibiotic Date & Time: | Antibiotic Date & Time: |
| | ECTION INFORMATION |
| Surgical Site Infection Type: | Culture Result: ☐ Positive ☐ Negative ☐ None taken |
| Superficial Incisional (up to 30 days only) | |
| Deep Incisional | Culture Date:(yyyy/mmm/dd)// |
| ☐ Organ-Space | Outline Torre (and managed) |
| Infection Onset Date: | Culture Type (see reverse): Organism isolated (if applicable): |
| | ☐ Coagulase negative <i>Staphylococcus</i> spp ☐ <i>Enterococcus</i> spp (specify): |
| yyyy/ | ☐ Staphylococcus aureus |
| yyyy/ miiiii / dd | ☐ Gram negative organism (specify): ☐ Other: |
| | Otali negative organism (specify). Other. |
| Clinical signs and symptoms of infection (check all that ap | poly): |
| Aseptically-obtained culture taken (fluid or tissue) | ☐ Dehiscence |
| Purulent drainage | ☐ Fever (>38°C) |
| Pain and/or tenderness | Incision deliberately opened by surgeon |
| Localized swelling, redness and/or heat | Abscess or other evidence of infection (on direct exam, during reoperation, by |
| ☐ Diagnosis of <b>superficial</b> SSI by surgeon, attending | histopathologic or radiologic examination) |
| physician or other designee | |
| Additional Infection Comments: | |
| CURREN | IT LOCATION INFORMATION |
| Re-admission Date: | Current Encounter Facility: |
| (if applicable) (yyyy/mmm/dd)// | - |
| Case Identification (check all that apply): | Current Encounter Zone: |
| Microbiology Report | Re-operation date (if applicable): |
| ☐ Emergency Room Visit | |
| Readmission to Hospital | |
| ☐ IV Antibiotic Therapy Clinic☐ Revision or other Surgical Procedure | yyyy/ mmm / dd |
| ☐ At Orthopaedic Surgeon Office | |
| ☐ At Orthopaedic Surgeon Office ☐ Observation of patient/incision/chart review | ICP Name: |
| Other (specify): | |

#### QUICK GUIDE FOR CDC/NHSN SURVEILLANCE DEFINTIONS (Feb. 2014)

1. Superficial incisional surgical site infection:

#### Infection occurs within 30 days after the operative procedure AND

Involves only skin and subcutaneous tissue of the incision AND

Patient has at least 1 of the following:

- a. Purulent drainage from the superficial incision.
- b. Organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision.
- c. Superficial incision that is **deliberately opened by a surgeon**, attending physician or other designee **and** is **culture positive or not cultured and** patient has **at least one of the following signs or symptoms**: pain or tenderness; localized swelling; redness; or heat. A culture negative finding does not meet this criterion.
- d. Diagnosis of a superficial incisional SSI by the surgeon or attending physician or other designee

#### 2. Deep incisional surgical site infection:

Infection occurs within 1 year if implant is in place and the infection appears to be related to the operative procedure AND Involves deep soft tissues (eq. fascia and muscle layers) of the incision AND

Patient has at least 1 of the following:

- a. Purulent drainage from the deep incision.
- b. A deep incision that spontaneously **dehisces** or is **deliberately opened by a** surgeon, attending physician or other designee **and** is **culture-positive or not cultured and** the patient has at least 1 of the following signs or symptoms: fever (>38°c); localized pain or tenderness. A culture-negative finding does not meet this criterion.
- c. An abscess or other evidence of infection involving the deep incision is found on direct examination, during reoperation, or by histopathologic or radiologic examination.

#### 3. Organ/space surgical site infection:

Infection occurs within 1 year if implant is in place and the infection appears to be related to the operative procedure AND Infection involves any part of the body, excluding the skin incision, fascia, or muscle layers, that is opened or manipulated during the operative procedure AND

Patient has at least 1 of the following:

- a. Purulent drainage from a drain that is placed through a stab wound into the organ/space.
- b. Organisms isolated from an **aseptically obtained culture** of fluid or tissue in the organ/space.
- C. An abscess or other evidence of infection involving the organ/space that is found on direct examination, during reoperation, or by histopathologic or radiologic examination and meets at least one criterion for a specific organ/space infection site listed in NHSN Table 4 here <a href="http://www.cdc.gov/nhsn/PDFs/pscManual/17pscNosInfDef">http://www.cdc.gov/nhsn/PDFs/pscManual/17pscNosInfDef</a> current.pdf

Table 4. Specific Sites of an Organ/Space SSI. Criteria for these sites can be found in the NHSN Help system (must be logged in to NHSN) or the Surveillance Definitions for Specific Types of Infections chapter.

| Code | Site | Code | Site |
|---|---|---|---|
| BONE | Osteomyelitis | LUNG | Other infections of the respiratory |
| | | | tract |
| BRST | Breast abscess or mastitis | MED | Mediastinitis |
| CARD | Myocarditis or pericarditis | MEN | Meningitis or ventriculitis |
| DISC | Disc space | ORAL | Oral cavity (mouth, tongue, or gums) |
| EAR | Ear, mastoid | OREP | Other infections of the male or female |
| | | | reproductive tract |
| EMET | Endometritis | OUTI | Other infections of the urinary tract |
| ENDO | Endocarditis | РЛ | Periprosthetic Joint Infection |
| EYE | Eye, other than conjunctivitis | SA | Spinal abscess without meningitis |
| GIT | GI tract | SINU | Sinusitis |
| HEP | Hepatitis | UR | Upper respiratory tract |
| IAB | Intraabdominal, not specified | VASC | Arterial or venous infection |
| IC | Intracranial, brain abscess or dura | VCUF | Vaginal cuff |
| JNT | Joint or bursa | | |

#### Culture Types: Fluid - aspirate Deep wound

Tissue

Superficial wound swab
Other

#### **Other Procedure Types:**

Misc. Surgery:

- Appendix
   Surgery
- Biliary Liver
- Pancreas
- Breast Surgery
- Colon Surgery
- Exploratory Abd Surgery
- Gallbladder Surgery
- Gastric Surgery
- Herniorrhaphy
- Kidney Surgery
- Neck Surgery
- Prostate Surgery
- Rectal Surgery
- Small Bowel Surgery
- Spleen Surgery
- Thoracic

#### OB-GYN:

- Abdominal Hysterectomy
- Caesarean Section
- Ovarian Surgery
- Vaginal Hysterectomy

#### Cardiac:

- CABG Chest Only
- CABG Chest and Donor
- Cardiac Surgery
- Pacemaker Surgery

#### Neurosurgery:

- Craniotomy
- Ventricular Shunt
- Laminectomy-Discectomy
- Spinal Fusion
- Spinal Re-fusion

#### Vascular:

- AAA Repair
- Atriovent Shunt Dialvsis
- Carotid Endarterectomy
- Vascular Bypass

#### Transplant:

- Heart Transplant
- Kidney Transplant
- Liver Transplant

### Local – Ortho:

- Limb Amputation
- Open Reduction
   Fracture
- Other Ortho Surgery
- Revision Hip
- Revision Knee

## **APPENDIX III: CASE REPORT FORMS**

| ELIGIBILITY AND ENROLLMENT | SWI-01 |
|----------------------------|--------|
| BASELINE CHARACTERISTICS | SWI-02 |
| INDEX SURGERY | SWI-03 |
| INDEX HOSPITAL DISCHARGE | SWI-04 |
| POSTOP LABORATORY RESULTS | SWI-05 |

| SW | VI-01: ELIGIBILITY AND ENROLLMENT PA | ATIENT ID: | |
|---|---|---|---|
| INC | LUSION CRITERIA: ALL RESPONSES MUST BE <u>YES</u> FOR ELIGIBILITY | | |
| 1. | Able to sign Informed Consent and Release of Medical Information Fo | orm □ Yes | □ No |
| 2. | Age ≥ 18 years | ☐ Yes | □ No |
| 3. | Undergoing cardiac surgery with complete sternotomy (including reoperations) | ☐ Yes | □ No |
| EXC | LUSION CRITERIA: ALL RESPONSES MUST BE <u>NO</u> FOR ELIGIBILITY | | |
| 1. | Evidence of active infection (any culture positive or blood positive inf | ection) 🗆 Yes | □ No |
| 2. | Undergoing organ transplantation | ☐ Yes | □ No |
| 3. | Known hypersensitivity to vancomycin | ☐ Yes | □ No |
| 4. | Pregnant or nursing women | ☐ Yes | □ No |
| 5. | Mental impairment or other conditions that may not allow participan understand the nature, significance, and scope of study | t to | □ No |
| Sigr | nature: — Date: — Date | DD/MMM/YYYY | |

07-May-2019 24

## SWI-02: BASELINE CHARACTERISTICS

| SW | 1-02: BASELINE CHARACTERISTICS | PATIENT ID: | |
|---|---|---|---|
| 1. | Last Name: | First Name: | |
| 2. | Date of birth (DD/MMM/YYYY): | / / | |
| 3. | PHN/ULI #: | | |
| 4. | Hospital ID#: | | |
| 5. | Walking | | |
| | ☐ No problems | | |
| 6. | Comments: | | ☐ Yes ☐ No |
| ь. | Immune deficiency Specify: | | ⊥ Yes ⊔ No |
| | Specify. | | |
| LAB | ORATORY PARAMETERS | | |
| Hen | natology Assessment Date (DD/MMM/Y | YYY): | |
| 1. | Hemoglobin (HGB) | □ □ □ g/L | |
| 2. | Hematocrit (HCT) | □.□□ L/L | |
| 3. | Platelet Count (PLT) | □ □ 10°/L | |
| 4. | White Blood Cell Count (WBC) | □. □ 10 <sup>9</sup> /L | |
| 5. | Neutrophil Count (NEUT) | □. □ 10 <sup>9</sup> /L | |
| 6. | Lymphocyte Count (LYMPH) | □. □ 10 <sup>9</sup> /L | |
| 7. | Monocyte Count (MONO) | □. □ 10 <sup>9</sup> /L | |
| 8. | Eosinophil Count (EOS) | □. □ 10 <sup>9</sup> /L | |
| 9. | Basophil Count (BASO) | □. □ 10 <sup>9</sup> /L | |
| Bloc | od Chemistry Assessment Date (DD/MN | им/үүүү): | |
| 10. | Sodium (Na) | □ □ □ mmol/L | |
| 11. | Potassium (K) | $\square$ . $\square$ mmol/L | |
| 12. | Urea | $\square$ . $\square$ mmol/L | |
| 13. | Creatinine (CR) | ☐ ☐ umol/L | |
| 14. | Glomerular filtration rate (GFR) | ☐ ☐ mL/min/1.73n | m² |

**2**5 07-May-2019

| Signature: Investigator/Coordinator | Date:DD/MMM/YYYY | _ |
|---|---|---|
| SWI-03: INDEX SURGERY | PATIENT ID: | |
| STUDY PRODUCT SYRINGE IDENTIFICATION N | UMBER: | |
| 1. Surgery date (DD/MMM/YYYY): | / | _ |
| 2. Was the chest closed in the OR? | ☐ Yes ☐ | No |
| ADVERSE REACTIONS TO STUDY PRODUCT | a along the sternal wound within 24 | No. |
| 1. Was there evidence of an allergic reaction hours of gauze application? | i along the sternal wound within 24 i res i | NO |
| DESCRIBE: | | |
| Signature: | Date: | |

## **SWI-04: INDEX HOSPITAL DISCHARGE**

| SW | /I-04: INDEX HOSPIT | AL DISCHARGE | | PATIENT ID: |
|-----|---------------------|--------------|-------|-------------|
| DIS | CHARGE ANTIBIOTIC | MEDICATIONS | | ☐ Yes ☐ No |
| | Cefazolin (ancef) | g | | |
| | Ciprofloxacin | mg | | |
| | Clindamycin | mg | | |
| | Flagyl | mg | | |
| | Gentamicin | mg/kg | | |
| | Vancomycin | g | | |
| | Other (specify): | | | |
| Sig | nature: | | Date: | DD/MMM/YYYY |

27 07-May-2019

| PATIENT ID: |
|-------------|

| ASSESSMENT | LABORATORY TEST | | | | | | |
|---|---|---|---|---|---|---|---|
| DATE AND TIME | CR | GFR | Urea Na K HGB | | | | HCT |
| DATE AND THISE | (umol/L) | (mL/min/1.73m <sup>2</sup> ) | (mmol/L) | (mmol/L) | (mmol/L) | (g/L) | (L/L) |
| | <u> </u> | | | | | 1 | |

| Signature: | | Date: - | |
|------------|--------------------------|---------|-------------|
| Signature. | Investigator/Coordinator | Date | DD/MMM/YYYY |

| PATIENT ID: |
|-------------|

| ASSESSMENT | LABORATORY TEST | | | | | | |
|---|---|---|---|---|---|---|---|
| DATE AND TIME | PLT<br>(10 <sup>9</sup> /L) | WBC<br>(10°/L) | NEUT<br>(10 <sup>9</sup> /L) | LYMPH<br>(10 <sup>9</sup> /L) | MONO<br>(10 <sup>9</sup> /L) | EOS<br>(10 <sup>9</sup> /L) | BASO<br>(10 <sup>9</sup> /L) |
| | , , | , , , | | | , , , | , , , | , , , |
| | l . | l . | l . | l . | l . | 1 | |

| Signature: | | Date: | |
|------------|--------------------------|-------|-------------|
| | Investigator/Coordinator | Date. | DD/MMM/YYYY |